CLINICAL TRIAL: NCT00483522
Title: The Effect of Scheduled Telephone Intervention on Outcomes After Traumatic Brain Injury
Brief Title: Telephone Intervention After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98-7055-C09
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Brain Injuries
Keywords: Rehabilitation; Directive counseling; Brain injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Scheduled telephone counseling over 2 years time.
  Interventions: Behavioral: Self-management telephone counseling
- 2 (No Intervention): This control group will receive standard care after hospital rehabilitation discharge as directed by their physician.

INTERVENTIONS:
Behavioral: Self-management telephone counseling — Subjects are contacted 7 times in year 1 after discharge from hospital rehabilitation unit and 4 times in year 2. Telephone counseling based on a self-management/problem-solving model is conducted by a research care manager.
  Arms: 1

SUMMARY:
This study seeks to determine if telephone counseling improves the outcome for persons with moderate to severe traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Subjects are recruited from the three participating TBI Model Systems of Care at Seattle, Philadelphia, and Jackson. After informed consent is obtained, some information is gathered about the injury and information about how the subject is doing cognitively, socially, and emotionally. After this information is obtained and after the subject is discharged from the acute rehabilitation unit, the subject is randomly selected to receive either standard care after discharge or standard care plus the telephone counseling.

The telephone follow-up group receives a telephone call from a research coordinator in 3-4 days, 2, 4, 8 weeks, and 5, 7, 9, 12, 15, 18, and 21 months after the date of injury. The research coordinator will work with the subject on problem-solving and self-management skills. In addition, the research coordinator will check in with a family member or friend for whom the subject has given permission to speak.

An outcome assessment is done by telephone at 12 months and 24 months after injury.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of traumatic brain injury upon admission to inpatient rehabilitation
* age 16 years or older
* arrival to an emergency department within 24 hours of acute injury
* receipt of both acute hospital care and inpatient rehabilitation within our facilities
* a permanent home address

Exclusion Criteria:

* previous hospitalization for TBI
* acute psychiatric disorder (e.g., schizophrenia or bipolar affective disorder)
* progressive neurological disease
* lack of a permanent home address
* discharge to a skilled nursing facility

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2004-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
A composite measure based on the measures of functional level, emotional status, community activities, and perceived quality of well-being. | One and two years

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Bell, M.D., Principal Investigator — University of Washington; Tessa Hart, Ph.D., Study Director — Moss Rehabilitation Research Institute; Mark Sherer, Ph.D., Study Director — Methodist Rehabilitation Center
Locations (3):
- United States (3):
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - Moss Rehabilitation Research Institute, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Bell KR, Esselman P, Garner MD, Doctor J, Bombardier C, Johnson K, Temkin N, Dikmen S. The use of a World Wide Web-based consultation site to provide support to telephone staff in a traumatic brain injury demonstration project. J Head Trauma Rehabil. 2003 Nov-Dec;18(6):504-11. doi: 10.1097/00001199-200311000-00004. PMID 14707880
- [Background] Bell KR, Hoffman JM, Doctor JN, Powell JM, Esselman P, Bombardier C, Fraser R, Dikmen S. Development of a telephone follow-up program for individuals following traumatic brain injury. J Head Trauma Rehabil. 2004 Nov-Dec;19(6):502-12. doi: 10.1097/00001199-200411000-00007. PMID 15602312
- [Background] Bell KR, Temkin NR, Esselman PC, Doctor JN, Bombardier CH, Fraser RT, Hoffman JM, Powell JM, Dikmen S. The effect of a scheduled telephone intervention on outcome after moderate to severe traumatic brain injury: a randomized trial. Arch Phys Med Rehabil. 2005 May;86(5):851-6. doi: 10.1016/j.apmr.2004.09.015. PMID 15895327
- [Background] Bell KR, Hoffman JM, Temkin NR, Powell JM, Fraser RT, Esselman PC, Barber JK, Dikmen S. The effect of telephone counselling on reducing post-traumatic symptoms after mild traumatic brain injury: a randomised trial. J Neurol Neurosurg Psychiatry. 2008 Nov;79(11):1275-81. doi: 10.1136/jnnp.2007.141762. Epub 2008 May 9. PMID 18469027
- [Background] Bombardier CH, Bell KR, Temkin NR, Fann JR, Hoffman J, Dikmen S. The efficacy of a scheduled telephone intervention for ameliorating depressive symptoms during the first year after traumatic brain injury. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):230-8. doi: 10.1097/HTR.0b013e3181ad65f0. PMID 19625862
- [Result] Hart T, Sherer M, Temkin N, Whyte J, Dikmen S, Heinemann AW, Bell K. Participant-proxy agreement on objective and subjective aspects of societal participation following traumatic brain injury. J Head Trauma Rehabil. 2010 Sep-Oct;25(5):339-48. doi: 10.1097/HTR.0b013e3181c7e60b. PMID 20042981
- [Result] Bell KR, Brockway JA, Hart T, Whyte J, Sherer M, Fraser RT, Temkin NR, Dikmen SS. Scheduled telephone intervention for traumatic brain injury: a multicenter randomized controlled trial. Arch Phys Med Rehabil. 2011 Oct;92(10):1552-60. doi: 10.1016/j.apmr.2011.05.018. PMID 21963122